CLINICAL TRIAL: NCT06577428
Title: Effect of Injection Site on the Relative Bioavailability of a Single Dose of RAY1225 in Subjects With Low and High Body Mass Index
Brief Title: A Study of RAY1225 at Different Injection Sites in Participants With Different Body Sizes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RAY1225-24-05
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RAY1225 - Upper Arm (Experimental): Participants received 3mg RAY1225 by subcutaneous injection on upper arm.
  Interventions: Drug: RAY1225
- RAY1225 - Thigh (Experimental): Participants received 3mg RAY1225 by subcutaneous injection on thigh.
  Interventions: Drug: RAY1225
- RAY1225 - Abdomen (Experimental): Participants received 3mg RAY1225 by subcutaneous injection on abdomen.
  Interventions: Drug: RAY1225

INTERVENTIONS:
Drug: RAY1225 — administered SC

SUMMARY:
The purpose of this study is to compare the amount of RAY1225 that gets into the blood stream and how long it takes the body to get rid of it, when injected under the skin of the upper arm and thigh compared to the abdomen. The study will be conducted in healthy males and females with different body sizes. The tolerability of RAY1225 will be evaluated and information about any side effects experienced will be collected. For each participant, the study will last about 7 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥19 kg/m2 and total body weight >50 kg for male, >45 kg for female at Screening (calculated as a function of measured height and weight according to the formula, BMI = kg / m2 where m2 is height in meters squared);
2. Ability to understand and willingness to sign a written informed consent form;
3. Normal physical examination, vital signs, 12-lead ECG, and clinical laboratory values, or any abnormality that is non-clinically significant.

Exclusion Criteria:

1. Participants with an allergic disposition (multiple drug and food allergies) or who, as determined by the investigator, are likely to be allergic to the investigational drug product or any component of the investigational drug product;
2. Participants had taken prescription, over-the-counter, herbal, or vitamin products within 14 days prior to screening；
3. Smoking more than 5 cigarettes per day within 3 months prior to screening，or who cannot stop using any tobacco products during the study period;
4. Participants who donated blood/bleeding profusely (> 400 mL) 3 months prior to randomization;
5. Those with clinically significant Electrocardiogram(ECG) abnormalities, or QTcF > 450ms;
6. Participants who test positive at screening for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), Hepatitis C virus (HCV) antibody or Syphilis spirochete-specific antibodies (TPPA);
7. Participants who test positive at Screening and/or admission (Day -1) for alcohol abuse.
8. Females who are pregnant, lactating, or likely to become pregnant during the study.
9. History of dysphagia or any gastrointestinal disorder that affect absorption;
10. Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve of RAY1225 From Time Zero to Infinity (AUC[0-∞]) | DAY1~43
PK: Maximum Concentration (Cmax) of RAY1225 | DAY1~43

SECONDARY OUTCOMES:
Number of participants with adverse events | DAY1~43

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Hospital of Chinese Medicine, Guanzhou, Guangdong, China